CLINICAL TRIAL: NCT00799734
Title: A Double-blind Randomized Placebo-controlled Clinical Trial on the Effects of Chinese Medicine Formula (Erxian Decoction) on Menopausal Symptoms
Brief Title: Chinese Medicine Therapy on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: School of Chinese Medicine, Li Ka Shing Faculty of Medicine, HKU, School of Chinese Medicine, HKU
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKCTR-740
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Menopause
Keywords: hot flushes; night sweats; menopausal symptoms; osteoporosis; complementary and alternative medicine
MeSH Terms: conditions — Hot Flashes; Osteoporosis | interventions — dixanthogen; er-xian decoction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alternative medicine (Active Comparator): Intake of prepacked Chinese herbal medicine (EXD), one sachet of granules (15g extracted granules) twice a day
  Interventions: Drug: EXD
- placebo (Placebo Comparator): placebo therapy of 15g granules with similar colour and taste.
  Interventions: Drug: EXD

INTERVENTIONS:
Drug: EXD — Interventions: Intake of prepacked Chinese herbal medicine therapy (EXD), one sachet of granules (15g extracted granules) twice a day and placebo therapy of 15g granules with similar colour and taste.
  Other Names: Er-xian Decoction (Prod. Code:3PP3082-3083)

SUMMARY:
The objective of this study is to evaluate whether a Chinese medicine formula (Erxian Decoction，EXD) is effective in alleviating menopausal symptoms, improving sex hormone profile and bone turn-over.

DETAILED DESCRIPTION:
This is a double-blind randomized placebo-controlled clinical trial to evaluate whether a Chinese medicine formula (Erxian Decoction) is effective in alleviating menopausal symptoms. This study will be conducted in Queen Mary Hospital and Chinese Medicine Clinic cum Training and Research Centers of the University of Hong Kong (Sassoon Road and Central). Women will be recruited from the general population by advertisements and promotion through media coverage.108 Chinese women with menopausal symptoms will be recruited and randomized into two groups.One is treatment group with 12 weeks of Erxian Decoction (well-controlled granules), the other is controlled group with 12 weeks of placebo. The treatment outcome measures include: 1) the severity of menopausal symptoms: self-recording of daily frequency of vasomotor symptoms (hot flushes plus night sweats),the Menopause-Specific Quality of Life (MENQOL) Questionnaire and the Menopause Rating Scale(MRS). 2)biochemical indices:serum follicle-stimulating hormone(FSH),luteinizing hormone(LH),estradiol, progesterone levels. 3)safety indices: blood count,liver and renal function tests. All measures are conducted at baseline and endpoint except the self-recoding of vasomotor symptoms and MENQOL Questionnaire, MRS. We expect this research will provide an effective and low-cost therapy for menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged 45 to 55 years old
2. having irregular menstrual cycles (≥3 months) indicating perimenopausal status or with cessation of menstrual period for at least three months within the previous 12 months
3. Total scores of Menopause Rating Scale≥28 indicating the menopausal symptoms are moderate or severe
4. Not having used HRT or Chinese Medicine for at least 3 months prior to entry into the study
5. Willing to give informed ,written consent to participate in the clinical study

Exclusion Criteria:

1. Taking hormones or medications, which could affect the vasomotoric symptoms
2. Having chronic illness, such as gastrointestinal, renal or liver disease, diabetes mellitus requiring treatment, uncontrolled hypertension
3. Having serious diseases, such as cancer, autoimmune system diseases, thrombosis and thrombophlebitis
4. Consuming alcohol, or taking psychiatric or psychotherapeutic drugs

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The severity of menopausal symptoms: self-recording of daily frequency of vasomotor symptoms (hot flushes plus night sweats),the Menopause-Specific Quality of Life (MENQOL) Questionnaire and the Menopause Rating Scale(MRS). | every four weeks

SECONDARY OUTCOMES:
bone markers (N-MID osteocalcin and serum crosslaps) | 12 weeks
Serum follicle-stimulating hormone (FSH), luteinizing hormone(LH), estradiol, progesterone levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yao Tong, PhD, Principal Investigator — School of Chinese Medicine, HKU
Locations (2):
- China (2):
  - Department of Obstetrics and Gynecology, the University of Hong Kong, Hong Kong, Hksar
  - Chinese Medicine Clinic cum Training and Research Centers of the University of Hong Kong, Hong Kong, Hong Kong